CLINICAL TRIAL: NCT04791501
Title: Prevalence and Outcome of Acute Hypoxemic Respiratory Failure in Children.
Brief Title: Prevalence AND Outcome of Acute Hypoxemic Respiratory fAilure in CHILDren (PANDORA-CHILD)
Acronym: PANDORA-child
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yolanda Lopez Fernandez (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Dr. Negrin University Hospital (Other)
Responsible Party: Sponsor-Investigator, Yolanda Lopez Fernandez, Principal Investigator, Hospital de Cruces
Organization: Hospital de Cruces (Other)
Other Study IDs: PI201935
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Respiratory Insufficiency
Keywords: respiratory failure; mechanical ventilation; children
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoxemic Respiratory Failure: Consecutive intubated patients receiving invasive mechanical ventilation with a PaO2/FiO2 ≤300 mmHg under a PEEP of 5 cmH2O or more and FiO2 of 0.3 or more.
  Interventions: Device: Mechanical ventilation

INTERVENTIONS:
Device: Mechanical ventilation — Ventilatory support

SUMMARY:
The present study is aimed to establish the epidemiological characteristics and clinical outcomes of mechanically ventilated children with acute hypoxemic respiratory failure (AHRF), defined as PaO2/FiO2 ≤300 mmHg on PEEP≥5 cmH2O and FiO2≥0.3, admitted in a network of pediatric hospitals in Spain.

DETAILED DESCRIPTION:
Prospective, multicenter, observational study focused on the prevalence and outcomes of Acute Hypoxemic Respiratory Failure in children. From a total of 40 pediatric ICUs in Spain, 22 PICUs agreed to participate.

All consecutive patients from 7 days to 16 years old admitted in the PICU will have been enrolled if they fulfilled the following criteria: 1) acute episode (within 7 days of a clinical insult), 2) on invasive mechanical ventilatory support, 3) PaO2/FiO2 ≤ 300 mmHg (or SpO2/FiO2 ≤ 264), 4) Positive end-expiratory pressure (PEEP) ≥ 5 cmH2O and FiO2 ≥ 0.3.

This study is considered an audit, and informed consent is waived.

Period of study: 2 years (October 2019 to September 2021). Recruitment period: two consecutive months (i.e October-November followed by a period of no recruitment) until complete 12 months of recruitment (September 2021).

All investigators have received guidelines outlining the study design and the methods for data collection. All PICU admissions are screened daily for AHRF. Onset of AHRF was defined as the day on which the patient first met all inclusion criteria. All data are collected on standardized forms. Demographics, comorbidities, reason for initiation of IMV, arterial blood gases, laboratory, radiographic, hemodynamic and ventilator data were collected at study entry and during the first three days of AHRF diagnosis (T0 or time of inclusion in the study, 24 hours, days 2 and 3). Chest imaging (chest radiographs, lung ultrasound or computed tomography) were evaluated daily for the presence or absence of infiltrates, atelectasis, acute pulmonary edema, pleural effusion or pneumothorax. Tidal volume (VT) was calculated on the basis of the predicted body weight (PBW). Plateau pressure (Pplat) was determined after the application of a 0.5- to 1.0-sec end-inspiratory hold. Driving pressure was calculated as the difference between Pplat and PEEP. Patients meeting pediatric ARDS criteria were stratified into a mild, moderate, and severe according to PALICC definition and/or berlin definition. All patients are followed until PICU and hospital discharge.

Data are initially collected and stored at each center and then sent to study coordinators at the time of patient's hospital discharge.

Although patient care is not strictly protocolized, physicians are asked to follow the current standards of pediatric critical care management. For ventilatory management, it was recommended that all patients be ventilated with a VT of 6-8 mL/kg PBW, at a ventilatory rate to maintain PaCO2 at 35-50 mm Hg, a Pplat <30 cm H2O, and PEEP and FiO2 combinations to maintain PaO2 >60 mm Hg or SpO2 >90%.

Statistical Analysis: for the main objective of the study, a descriptive analysis including clinical variables, mechanical ventilation data, respiratory settings and ancillary measures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 7 days to 16 years old admitted in the PICU.
* Acute episode (within 7 days of a clinical insult)
* On invasive mechanical ventilatory support
* PaO2/FiO2 ≤ 300 mmHg (or SpO2/FiO2 ≤ 264)
* Positive end-expiratory pressure (PEEP) ≥ 5 cmH2O and FiO2 ≥ 0.3.

Exclusion Criteria:

* Non-invasive respiratory support *Aged >16 years or < 7 days.

Ages: 7 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive patients from 7 days to 16 years old admitted in the PICU with an acute episode (within 7 days of a clinical insult) of hipoxemia defined as PaO2/FiO2 ≤ 300 mmHg (or SpO2/FiO2 ≤ 264), and on invasive mechaniccal ventilatio with a PEEP ≥ 5 cmH2O and FiO2 ≥ 0.3.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypoxemic acute respiratory failure. | 12 months
  The investigators will calculate the prevalence in relation to: (i) total number of ICU admissions during the study period in all participating centers; (ii) total number of mechanically ventilated patients during the study period in all participating centers, and (iii) per ICU bed available in the participating centers over the study period.

SECONDARY OUTCOMES:
Death in the ICU and in the hospital | through study completion, an average of 60 days
  Outcome after discharge from ICU and before discharge to home (overall and in each category of acute hypoxemic respiratory failure).

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar Hernández, MD, PhD, Study Director — Multidisciplinary Organ Dysfunction Evaluation Research Network (MODERN). Research Unit, hospital universitario dr. negrín, Las Palmas de gran Canaria, Spain.
Locations (23):
- Spain (23):
  - Cruces University Hospital, Barakaldo, Bizkaia
  - Complejo Hospitalario Donosti, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Madrid
  - Niño Jesús University Hospital, Madrid
  - Hospital Universitario, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Camino, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen de la Salud, Toledo
  - Hospital Universitario La fe, Valencia
  - Hospital Clinico Universitario, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Fernandez Y, Azagra AM, de la Oliva P, Modesto V, Sanchez JI, Parrilla J, Arroyo MJ, Reyes SB, Pons-Odena M, Lopez-Herce J, Fernandez RL, Kacmarek RM, Villar J; Pediatric Acute Lung Injury Epidemiology and Natural History (PED-ALIEN) Network. Pediatric Acute Lung Injury Epidemiology and Natural History study: Incidence and outcome of the acute respiratory distress syndrome in children. Crit Care Med. 2012 Dec;40(12):3238-45. doi: 10.1097/CCM.0b013e318260caa3. PMID 22990455
- [Background] Villar J, Blanco J, Anon JM, Santos-Bouza A, Blanch L, Ambros A, Gandia F, Carriedo D, Mosteiro F, Basaldua S, Fernandez RL, Kacmarek RM; ALIEN Network. The ALIEN study: incidence and outcome of acute respiratory distress syndrome in the era of lung protective ventilation. Intensive Care Med. 2011 Dec;37(12):1932-41. doi: 10.1007/s00134-011-2380-4. Epub 2011 Oct 14. PMID 21997128
- [Background] Kopczynska M, Sharif B, Pugh R, Otahal I, Havalda P, Groblewski W, Lynch C, George D, Sutherland J, Pandey M, Jones P, Murdoch M, Hatalyak A, Jones R, Kacmarek RM, Villar J, Szakmany T, On Behalf Of The Pandora-Wales Investigators. Prevalence and Outcomes of Acute Hypoxaemic Respiratory Failure in Wales: The PANDORA-WALES Study. J Clin Med. 2020 Oct 31;9(11):3521. doi: 10.3390/jcm9113521. PMID 33142837
- [Derived] Lopez-Fernandez YM, Martinez-de-Azagra A, Reyes-Dominguez SB, Gomez-Zamora A, Herrera-Castillo L, Coca-Perez A, Parrilla-Parrilla J, Medina A, Garcia-Iniguez JP, Brezmes-Raposo M, Hernandez-Yuste A, Llorente de la Fuente AM, Ibarra de la Rosa I, Leon-Gonzalez JS, Trastoy-Quintela J, Arjona-Villanueva D, Gonzalez-Martin JM, Szakmany T, Villar J; Prevalence AND Outcome of acute hypoxemic Respiratory fAilure in children (PANDORA-CHILD) Network. The Prevalence and Outcome of Acute Hypoxemic Respiratory Failure (PANDORA) Study in Mechanically Ventilated Children: Prospective Multicenter Epidemiology in Spain, 2019-2021. Pediatr Crit Care Med. 2025 Jun 1;26(6):e759-e772. doi: 10.1097/PCC.0000000000003743. Epub 2025 Apr 25. PMID 40277417